CLINICAL TRIAL: NCT00081783
Title: A Phase II Study of Xcellerated T CellsTM in Patients With Relapsed or Refractory Indolent Non-Hodgkin's Lymphoma (NHL)
Brief Title: Xcellerated T CellsTM for Non-Hodgkin's Lymphoma (NHL) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xcyte Therapies (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XT009
Record Dates: First submitted 2004-04-20; First posted 2004-04-22 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-03

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: T Cells; Immunotherapy; NHL; Xcellerated T Cells
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

INTERVENTIONS:
Drug: Xcellerated T Cells

SUMMARY:
This is a Phase II single arm study of a novel T cell immunotherapy in patients with indolent non-Hodgkin's lymphoma (NHL). Eligible patients will have relapsed or refractory disease after receiving at least one and no more than four prior regimens. Patients will receive Xcellerated T CellsTM, an ex vivo activated and expanded autologous T cell product, in an attempt to enhance immune responses with anti-tumor activity. The primary endpoint of the study is to evaluate the efficacy of Xcellerated T Cells in patients with indolent NHL. Secondary endpoints are to evaluate the safety of the therapy in this patient population, and to evaluate changes in the number and phenotype of T- and B-lymphocytes, as well as changes in the T cell receptor repertoire, hemoglobin levels, platelet counts and quantitative immunoglobulin levels. In a subset of patients, fine-needle aspirates of malignant lymph nodes will be performed to assess changes in the lymphocyte composition and phenotype. Bone marrow aspirates will be similarly evaluated. Finally, anti-tumor immune responses will be evaluated in patients amenable to biopsy of enlarged lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Indolent non-Hodgkin's Lymphoma (NHL), with one of the following subtypes according to the REAL Classification: follicular lymphoma, small lymphocytic lymphoma (SLL), extranodal marginal zone B-cell lymphoma (MALT), nodal marginal zone B-cell lymphoma (monocytoid B-cell lymphoma), splenic marginal zone lymphoma (splenic lymphoma with villous lymphocytes) and mantle cell lymphoma. Other subtypes require approval of the Medical Monitor. At least 16 patients with small lymphocytic lymphoma, and no more than eight patients with mantle cell lymphoma will be enrolled.
* Stage III or IV disease at any time in the past
* Relapsed or refractory disease following most recent treatment. Patients are considered to have refractory disease if their last treatment course did not result in a complete or partial response, or if time to disease progression was six months or less. Patients are considered to have relapsed disease if time to disease progression is more than six months. Patients who have achieved a partial or complete response following most recent therapy must have demonstrated progressive disease.
* Patients must have received at least one prior course of systemic therapy for NHL and no more than four prior courses of therapy. Repeat courses of the same therapeutic regimen separated in time by six or more months are considered separate treatment courses, with the exception of single-agent rituximab. Patients with more than four prior courses of therapy may be enrolled at the discretion of the Medical Monitor after discussion with the Investigator.
* Radiographically bi-dimensionally measurable disease. Imaging need not be performed within 15 days prior to registration. Prior scans are acceptable provided that there has been no intervening therapy for NHL. Scans will be obtained at baseline, following registration.
* Age of at least 18 years
* ECOG performance status of 0 to 2
* White blood count (WBC) ≥ 3,000/mm3, absolute neutrophil count (ANC) ≥ 1000/mm3
* CD3+ > 1% of total peripheral white blood cell count by flow cytometry
* Platelet count > 50,000/mm3
* Hemoglobin ³ 10.0 g/dL. Transfusion with red blood cells or use of erythropoietin is permissible.
* Serum total bilirubin and alanine aminotransferase (ALT) ≤ 2.0 times the upper limit of normal
* Serum creatinine ≤ 2.0 mg/dL
* Serum human anti-mouse antibody (HAMA) titer undetectable or within the normal range, and no history of symptomatic allergic reactions to mice or murine (mouse) proteins. Patients with elevated HAMA levels may be enrolled at the discretion of the Medical Monitor after discussion with the Investigator.
* Negative test results for current/active infection with HIV-1, HIV-2, HTLV-1, HTLV-2, hepatitis B and hepatitis C within 30 days of registration. (Antibody, antigen and nucleic acid tests acceptable, depending on institutional standards)
* Women of childbearing potential must have a negative serum pregnancy test. Both men and women agree to use a medically accepted form of contraception from the time of initial screening through completion of the study.
* Able to comprehend and provide signed informed consent

Exclusion Criteria:

* Evidence of Hodgkin's lymphoma, Burkitt's lymphoma, diffuse large B-cell lymphoma, primary mediastinal B-cell lymphoma, lymphoplasmacytic lymphoma, hairy cell leukemia, primary central nervous system lymphoma or any other aggressive lymphoma
* Any T cell lymphoma
* Evidence of primary cutaneous anaplastic large cell lymphoma, Richter's Syndrome, large granular lymphocytosis and Sézary-cell leukemia. Patients with a prior diagnosis of chronic lymphocytic leukemia, as evidenced by absolute peripheral lymphocyte count of greater than 5,000 per mm3 at any time in the past, are not eligible.
* Leukemic manifestations of non-Hodgkin's lymphoma. Small lymphocytic lymphoma patients with peripheral lymphocyte count greater than 5,000 per mm3
* Receipt of any chemotherapy, monoclonal antibody, investigational or other systemic therapy (except glucocorticoids as noted below) for the treatment of NHL within 2 months prior to registration
* Receipt of glucocorticoids (with the exception of inhaled glucocorticoids) within 1 month prior to registration
* Receipt of intravenous immunoglobulin (IVIG) within 1 month of registration
* Registration for, or plans to participate in, any other clinical trial of an investigational agent concurrently with this trial
* History of malignancy other than NHL within five years of registration, except adequately treated basal or squamous cell skin cancer or in situ carcinoma of the cervix. Other exceptions must be approved by the Xcyte Therapies' Medical Monitor prior to registration.
* Infection requiring treatment with antibiotics, antifungal, or antiviral agents within seven days of registration
* Active autoimmune disease requiring systemic treatment
* Major organ system dysfunction including (but not limited to): New York Heart Association Class III or IV, severe pulmonary, renal, hepatic, gastrointestinal, neurologic or psychiatric dysfunction which would impair patient's ability to participate in the trial
* Any other pertinent medical or psychological condition which leads the Investigator to believe the study would not be appropriate treatment or in the patient's best interest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: Mark W. Frohlich, MD, Study Chair — Xcyte Therapies
Locations (18):
- United States (18):
  - California Cancer Care, Greenbrae, California
  - University of Southern California, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Atlanta Cancer Care, Roswell, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Center for Cancer & Blood Disorders, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ohio State University, Columbus, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Virginia Mason, Seattle, Washington